CLINICAL TRIAL: NCT04450966
Title: Computer-facilitated Screening and Brief Intervention (cSBI) in Pediatric Primary Care to Reduce Underage Drinking: a Large, Multi-site Randomized Trial
Brief Title: Adolescent Substance Use Prevention Intervention Research Study in Pediatric Primary Care
Acronym: ASPIRE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: American Academy of Pediatrics (Other); Children's Hospital of Philadelphia (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Sion Kim Harris, Associate Professor of Pediatrics, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIAAA_1R01AA027253-01A1
Record Dates: First submitted 2020-06-25; First posted 2020-06-30 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-01

CONDITIONS: Heavy Drinking; Driving Under the Influence; Riding With Driver Under the Influence
MeSH Terms: conditions — Driving Under the Influence | interventions — Crisis Intervention

STUDY DESIGN:
Intervention Model Description: Multi-site cluster-randomized parallel groups trial. >30 pediatric primary care clinicians will be recruited from ~10 practices and will be allocated 1:1 to either deliver usual care or the cSBI intervention to their participating patients ages 14-17 years-old.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (No Intervention): Clinicians randomized to this arm will not receive training in delivery of cSBI until study completion, and their participating patients will receive usual care.
- Computer-facilitated screening and brief intervention (Experimental): Clinicians randomized to this arm will receive training in delivery of cSBI and their participating patients will then receive the experimental intervention.
  Interventions: Behavioral: Computer-facilitated Screening and Brief Intervention

INTERVENTIONS:
Behavioral: Computer-facilitated Screening and Brief Intervention — cSBI includes: 1) computer self-administered screening that adolescents complete prior to seeing their clinician, immediately followed by 2) computer-delivered brief psychoeducation on the health risks of substance use to prime patients for the clinician encounter, and 3) a Clinician Report Form with screen results and prompts that clinicians use to provide motivational interviewing-based individualized counseling during the visit.
  Other Names: cSBI
  Arms: Computer-facilitated screening and brief intervention

SUMMARY:
Our goal is to conduct a large multi-site randomized controlled trial (RCT) of a promising computer-facilitated Screening and clinician Brief Intervention (cSBI) system designed for delivery by pediatric primary care clinicians and aimed at reducing unhealthy alcohol use and related riding/driving safety risk among adolescent patients. Our setting will be the American Academy of Pediatrics' (AAP) Pediatric Research in Office Settings (PROS) national primary care research network, with >600 U.S. primary care practices having participated in recent studies. This trial addresses the evidence gap identified in the latest U.S. Preventive Services Task Force review of alcohol screening and brief counseling interventions among adolescents, and, if shown effective, the cSBI system could be widely disseminated via AAP's existing education, teaching, and advocacy platforms to its 67,000 pediatrician members, thereby greatly increasing the potential for population-level impact of alcohol screening and brief intervention for U.S. adolescents.

DETAILED DESCRIPTION:
Alcohol use disorders frequently have a pediatric origin. Pediatric primary care offices, where the majority of adolescents receive health care, are a promising venue for early identification and intervention through universal screening and brief counseling. However, while the U.S. Preventive Services Task Force recommends primary care-based alcohol screening and brief intervention for adults, it found insufficient evidence to recommend it for adolescents.

The goal of the proposed study is to address this evidence gap by testing the effectiveness of a promising computer-facilitated Screening and Brief Intervention (cSBI) system for delivery by pediatric primary care clinicians to adolescents at well-visits. This cluster-randomized controlled trial will be conducted in the American Academy of Pediatrics' (AAP) Pediatric Research in Office Settings (PROS) national primary care practice-based research network. PROS has demonstrated success in >30 years of practice-based research, with >600 practices participating in recent studies. Drawing on more than 15 years of our prior research on adolescent alcohol screening and brief counseling in primary care offices, the cSBI system was developed to provide a time-efficient and feasible way for pediatric practices to improve both the frequency and quality of alcohol screening and counseling. cSBI includes: 1) computer self-administered screening that adolescents complete prior to seeing their clinician, 2) 10 interactive psychoeducational pages for the adolescent on substance use health risks, 3) a Clinician Report Form with screen results and prompts that clinicians use to provide motivational interviewing-based individualized counseling, and 4) clinician training materials and protocol.

In a New England-based pilot study, we found that, compared to usual care (UC), the cSBI approach: 1) increased patient receipt of alcohol-related counseling during well-visits; 2) improved patients' ratings of the quality of their clinician encounter; and 3) among those who reported past-year use at baseline (n=192), was associated with a 34% lower risk of a heavy episodic drinking episode during 12 months follow-up. cSBI also reduced risk of riding with an impaired driver, a major safety risk associated with alcohol, by 42% among those with prior riding risk.

A larger RCT of this approach, which employs an adequately-powered sample and tests generalizability of effects beyond New England, is needed. We will randomize >30 pediatric primary care clinicians in ~10 practices nationwide to deliver UC or cSBI (1:1) to their eligible and assenting 14- to 17-year-old patients arriving for well-visits. Our aims are to test cSBI's effect on adolescent patients' heavy episodic drinking, and on riding with an impaired driver/driving while impaired, during 12 months follow-up. We hypothesize that, compared to adolescent patients receiving usual care, those receiving cSBI will have lower rates of reporting heavy episodic drinking and riding with an impaired driver/driving while impaired during the study follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Ages 14-17
* Presenting for well-visit with participating clinician
* Reports any lifetime alcohol use
* If no lifetime alcohol use, reports riding with a driver under the influence in the past 12 months
* Has own cell phone and is willing to share cell phone number before their scheduled visit
* Completes required pre-visit activity/activities before well visit

Exclusion Criteria:

* Youth in foster care
* Unable to read and communicate in English
* Unable to complete follow-ups
* Currently receiving treatment from specialty clinician(s) for a substance use concern
* Deemed by their clinician to be inappropriate for study participation due to neurodevelopmental delays or medical/emotional concerns

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 406 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Any heavy episodic drinking day during past 3 months | 3 months follow-up
  Defined using the NIAAA Youth Guide age/gender-specific number of drinks.
Any heavy episodic drinking day during past 3 months | 6 months follow-up
  Defined using the NIAAA Youth Guide age/gender-specific number of drinks.
Any heavy episodic drinking day during past 3 months | 9 months follow-up
  Defined using the NIAAA Youth Guide age/gender-specific number of drinks.
Any heavy episodic drinking day during past 3 months | 12 months follow-up
  Defined using the NIAAA Youth Guide age/gender-specific number of drinks.
Time to first day of heavy episodic drinking during 12 month follow-up period | 1-12 months follow-up
  Deﬁned using the NIAAA Youth Guide age/gender- speciﬁc number of drinks.

SECONDARY OUTCOMES:
Any riding/driving risk | 3 months follow-up
  Any riding with a driver who had been using alcohol or driving after using alcohol in past 3 months
Any riding/driving risk | 6 months follow-up
  Any riding with a driver who had been using alcohol or driving after using alcohol in past 3 months
Any riding/driving risk | 9 months follow-up
  Any riding with a driver who had been using alcohol or driving after using alcohol in past 3 months
Any riding/driving risk | 12 months follow-up
  Any riding with a driver who had been using alcohol or driving after using alcohol in past 3 months

OTHER OUTCOMES:
Alcohol-related problems or negative consequences experienced since post-visit survey | 6 months follow-up
  Score on scale
Alcohol-related problems or negative consequences experienced since post-visit survey | 12 months follow-up
  Score on scale
Past 3 months alcohol use days | 3 months follow-up
  Number of days of any alcohol use in past 3 months
Past 3 months alcohol use days | 6 months follow-up
  Number of days of any alcohol use in past 3 months
Past 3 months alcohol use days | 9 months follow-up
  Number of days of any alcohol use in past 3 months
Past 3 months alcohol use days | 12 months follow-up
  Number of days of any alcohol use in past 3 months
Past 3 months heavy episodic drinking days | 3 months follow-up
  Number of days of heavy episodic drinking in past 3 months
Past 3 months heavy episodic drinking days | 6 months follow-up
  Number of days of heavy episodic drinking in past 3 months
Past 3 months heavy episodic drinking days | 9 months follow-up
  Number of days of heavy episodic drinking in past 3 months
Past 3 months heavy episodic drinking days | 12 months follow-up
  Number of days of heavy episodic drinking in past 3 months
Perceived risk of harm | 3 months follow-up
  Percent report perceiving moderate/great risk of harm from regular heavy episodic drinking
Perceived risk of harm | 6 months follow-up
  Percent report perceiving moderate/great risk of harm from regular heavy episodic drinking
Perceived risk of harm | 12 months follow-up
  Percent report perceiving moderate/great risk of harm from regular heavy episodic drinking
Drinking refusal self-efficacy | 3 months follow-up
  Score on Drinking Refusal Self-Efficacy measure
Drinking refusal self-efficacy | 6 months follow-up
  Score on Drinking Refusal Self-Efficacy measure
Drinking refusal self-efficacy | 12 months follow-up
  Score on Drinking Refusal Self-Efficacy measure

CONTACTS AND LOCATIONS:
Overall Officials: Sion K Harris, PhD, Principal Investigator — Boston Children's Hospital; Lydia A Shrier, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (3):
- United States (3):
  - American Academy of Pediatrics, Itasca, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
We will provide a variable codebook along with the dataset. We will make a de-identified version of the complete and cleaned study dataset available to the AAP's PROS Study Archive at study completion, as well as NIAAA Data Archive (NIAAADA).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 12 months of study completion.
Access Criteria: We will share the dataset with external investigators when a data use agreement (DUA) is executed between Boston Children's Hospital and the institution of the person making the request. The DUA will specify the requested data elements (each of which must be justified), the specific research question, the timeline for the project and schedule for data destruction.

REFERENCES:
- [Derived] Shrier LA, O'Connell MM, Torres A, Shone LP, Fiks AG, Plumb JA, Maturo JL, McCaskill NH, Harris D, Burke PJ, Felt T, Murphy ML, Sherritt L, Harris SK. Computer-Facilitated Screening and Brief Intervention for Alcohol Use Risk in Adolescent Patients of Pediatric Primary Care Offices: Protocol for a Cluster Randomized Controlled Trial. JMIR Res Protoc. 2024 Mar 26;13:e55039. doi: 10.2196/55039. PMID 38530346